CLINICAL TRIAL: NCT02439086
Title: Prediction of Response to Neoadjuvant Chemoradiotherapy in Locally Advanced Rectal Cancer.
Brief Title: Prediction of Response to Neoadjuvant Therapy in Rectal Cancer
Acronym: PRENT-LARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Colchester General Hospital (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Principal Investigator, Medhat Alaker, Principal Investigator, Colchester General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: TBA (ethics)
Record Dates: First submitted 2015-04-23; First posted 2015-05-08 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Rectal Neoplasms
Keywords: rectal cancer; neoadjuvant chemoradiotherapy; long course radiotherapy; response
MeSH Terms: conditions — Rectal Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Long Course Radiotherapy (Experimental): all patients diagnosed with rectal cancer, amenable for neoadjuvant chemoradiotherapy, who agree to participate in this study will undergo 2 PET-CT scans: at baseline and 9 weeks after commencing therapy.
  Interventions: Device: PET-CT Scan

INTERVENTIONS:
Device: PET-CT Scan — patients will have 2 PET CT scans: one before radiotherapy, and one 9 weeks after.

SUMMARY:
The purpose of this study is to determine whether 18F-FDG-PET-CT and texture analysis of MRI performed 9 weeks after Neoadjuvant Chemo-radiotherapy in patients with locally advanced rectal cancer has the ability to identify patients with Complete Response.

DETAILED DESCRIPTION:
In recent years, treatment with NCRT has revolutionised management of LARC. In addition to downstaging the tumour in 62% of cases, half of which decrease by more than 1 T stage; pathological complete response (pCR), with no viable tumour cells left in resected specimens, was demonstrated in up to 30% of patients. Only 3% of patients showed progressive disease. It has recently been shown that those with pathological complete response survive longer than those with partial response, with figures for 5-year disease free survival quoted between 83 and 91% for pCR; versus 65% for non pCR. Furthermore, it has been argued that those tumours which are sensitive to radiotherapy have a favourable biological tumour profile, with fewer propensities to recur or to metastasise than aggressive non-radiosensitive tumours. The key is to accurately be able to identify patients who exhibit complete response to radiotherapy, or to predict those who might show complete response.

Positron Emission Tomography (18-F-FDG-PET-CT) as a tumour biomarker after radiotherapy has been shown to be able to predict patients who have responded to chemo radiotherapy, with a sensitivity of 79% and specificity of 88%. Texture Analysis (TA) assesses the aggressiveness of the tumour by assessing intra-tumoural heterogeneity. It has already been shown to be effective in assessing biological characteristics of solid tumours, including the oesophagus, breast, and liver.

The aim of this study is to utilise these two novel molecular imaging techniques to identify rectal cancer patients who have responded completely from neoadjuvant chemo-radiotherapy. Parameters will be calculated as changes in measurable variables from baseline to post treatment scans.

Pilot data The watch-and-wait approach could potentially reduce treatment-related toxicity in selected rectal cancer patients who have a clinical complete response (cCR) after chemoradiation. The "watch & wait" protocol has been adopted from studies performed in Brazil, United Kingdom, and the Netherlands.

Studies indicate that accurate assessment of response to neoadjuvant therapy is the key to selecting patients who will benefit from the watch & wait approach. Therefore, determining the modality with highest accuracy and cost-effectiveness has been the holy grail of managing locally advanced rectal cancers.

A study performed by our Chief Investigator on the efficiency and accuracy of 18-F-FDG-PET-CT has concluded that PET-CT has a proven role and is cost effective in monitoring therapy and in detecting recurrence in colorectal cancers; as this technology combines picomolar sensitivity with high-resolution CT imaging. It has therefore shown to be more sensitive than plain CT imaging in detecting recurrence and monitoring response to therapy. In other studies, the reported accuracy for PET-CT in determining responsiveness to NCRT was around 80%. Baseline PET-CT and subsequent PET-CT parameters, including SUV-based measurements, have been shown to be highly accurate in determining responses to NCRT.

Texture Analysis is a biomarker technique that measures heterogeneity within solid tumours. Textural parameters (coefficient of variation [COV], skewness, and kurtosis) applied on PET-CT images has been shown to be able to predict response to NCRT, and to predict survival. A pilot study performed at our institution has indeed showed that textural parameters performed on pelvic MRI were associated with improved overall survival and disease- free survival.

Study hypothesis

* PET-CT restaging done at 9 weeks rather than 6 weeks will be a more accurate predictor in assessing response to NCRT.
* Texture analysis of rectal MRI scans is a strong biomarker in assessing tumour response and identifying patients with Complete Response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven confirmed rectal cancer
* MRI stage: T3/T4 and/or N1/N0.
* No contraindication to MRI and PET-CT.

Exclusion Criteria:

* Contraindication to MRI and/or PET-CT.
* Inability to consent.
* Severe claustrophobia.
* Distant metastases.
* Synchronous tumour.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Texture analysis PET-CT | 6 months
  Sensitivity will be calculated from 2x2 contingency table.

SECONDARY OUTCOMES:
Correlation between tumour response parameters to survival. | 6 months
  Correlation coefficient (r)
Accuracy of Texture analysis MRI | 6 months
  Sensitivity will be calculated from 2x2 contingency table.

CONTACTS AND LOCATIONS:
Overall Officials: Tan Arulampalam, MD, Principal Investigator — ICENI Centre director
Locations (1):
- Colchester General Hospital, Colchester, United Kingdom

REFERENCES:
- [Background] Arulampalam TH, Costa DC, Loizidou M, Visvikis D, Ell PJ, Taylor I. Positron emission tomography and colorectal cancer. Br J Surg. 2001 Feb;88(2):176-89. doi: 10.1046/j.1365-2168.2001.01657.x. PMID 11167864
- [Background] Bundschuh RA, Dinges J, Neumann L, Seyfried M, Zsoter N, Papp L, Rosenberg R, Becker K, Astner ST, Henninger M, Herrmann K, Ziegler SI, Schwaiger M, Essler M. Textural Parameters of Tumor Heterogeneity in (1)(8)F-FDG PET/CT for Therapy Response Assessment and Prognosis in Patients with Locally Advanced Rectal Cancer. J Nucl Med. 2014 Jun;55(6):891-7. doi: 10.2967/jnumed.113.127340. Epub 2014 Apr 21. PMID 24752672
- [Background] HABR-GAMA, A., PEREZ, R., LYNN, P., SÃ£O JULIÃ£O, G. and GAMA RODRIGUES, J., 2012. Selective non-operative management of distal rectal cancer: The Watch & Wait Protocol. In: R. SCHIESSEL and P. METZGER, eds, Springer Vienna, pp. 43-53.
- [Background] Habr-Gama A, Perez RO, Nadalin W, Sabbaga J, Ribeiro U Jr, Silva e Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Operative versus nonoperative treatment for stage 0 distal rectal cancer following chemoradiation therapy: long-term results. Ann Surg. 2004 Oct;240(4):711-7; discussion 717-8. doi: 10.1097/01.sla.0000141194.27992.32. PMID 15383798
- [Background] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Background] Niccoli-Asabella A, Altini C, De Luca R, Fanelli M, Rubini D, Caliandro C, Montemurro S, Rubini G. Prospective analysis of 18F-FDG PET/CT predictive value in patients with low rectal cancer treated with neoadjuvant chemoradiotherapy and conservative surgery. Biomed Res Int. 2014;2014:952843. doi: 10.1155/2014/952843. Epub 2014 May 4. PMID 24877151
- [Derived] Aker M, Ganeshan B, Afaq A, Wan S, Groves AM, Arulampalam T. Magnetic Resonance Texture Analysis in Identifying Complete Pathological Response to Neoadjuvant Treatment in Locally Advanced Rectal Cancer. Dis Colon Rectum. 2019 Feb;62(2):163-170. doi: 10.1097/DCR.0000000000001224. PMID 30451764